CLINICAL TRIAL: NCT06365268
Title: Perinatal Thoraco-abdominal Tumors Management in Infants : a Multicenter Experience
Brief Title: Perinatal Thoraco-abdomino-pelvic Tumors Study
Acronym: CONTRAST
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231139
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Solid Tumors of the Thoraco-abdomino-pelvic Region
Keywords: Congenital truncal tumors; Antenatal diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Mother-child whose care course for the child's congenital axial tumor included treatment at the AP-HP between 2010 and 2021. Fetus presenting a malignant or benign solid tumor of thoracic, abdominal or pelvic location and whose clinico-radiological or histological diagnosis is confirmed postnatally up to 1 year of life with the onset of symptoms in the first three months of life.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file. The data collected concerns a period of three years maximum.

SUMMARY:
Congenital tumors are a rare diagnosis in the fetus and newborn. They differ from those of children and adults in terms of the nature, location and evolution of the tumor.

Indeed, some histologically benign tumors may have lethal potential in utero (e.g. sacrococcygeal teratomas) or even undergo malignant transformation if left untreated. In contrast, other tumors that are malignant by histological criteria may have a very good prognosis, regressing spontaneously within the first year of life (e.g. neuroblastoma).

Despite advances in imaging, benign and malignant solid tumors remain a major diagnostic and prognostic challenge in the antenatal context.

The management of congenital tumors requires multidisciplinary expertise, taking into account the perinatal context, which poses specific problems, particularly in terms of therapeutic aspects, but also the frequent existence of associated malformations and/or genetic predisposition syndromes.

This study focuses on solid tumors of the thoraco-abdomino-pelvic region, the main objective being to investigate the correlation between antenatal clinical and radiological analysis and confirmed postnatal diagnosis of congenital solid truncal tumors, as well as the developmental spectrum in which they fit.

DETAILED DESCRIPTION:
Congenital tumors are a rare diagnosis in the fetus and newborn. Despite advances in imaging techniques, it remains a major diagnostic and prognostic challenge. The congenital tumor differs from that of the child and adult in terms of tumoral nature, localization and evolution.

The investigation of a congenital tumor must be multidisciplinary and exhaustive, since it is estimated that congenital tumors are associated with a genetic predisposition syndrome in 10% to 15% of cases, and this proportion is set to rise in the coming years.

Precise analysis of the spectrum of tumors involved, and diagnosis of the nature of the tumor, are the basis for advice and pre- and post-natal care. Prenatal information given to parents must be accurate and precise, as the diagnosis of a congenital tumor may lead to a request for medical termination of pregnancy.

Diagnostic performance in the characterization of a tumor mass in antenatal care is still imperfect.

Diagnostic performance in the characterization of a tumor mass in antenatal care is still imperfect.

By reporting on our experience in the management of congenital tumors in the Ile-de-France region, we aim to improve our understanding of the developmental spectrum in which these tumors occur. By clarifying the diagnosis, the resulting management can be optimized and adapted to each situation. The challenge is to treat the tumor effectively and sustainably, while avoiding overly aggressive treatments when they are not indicated. Post-natal therapies will be described in detail for each situation, to produce a simplified algorithm for management.

The quality of this information will condition the parents' experience and avoid requests for medical termination of pregnancy for benign tumors and/or spontaneous involution. On the contrary, this will be discussed in rare cases of very aggressive tumor involving the functional or vital prognosis of the unborn child or occurring in a context of known genetic predisposition.

ELIGIBILITY:
Inclusion Criteria:

* Information of the holders of parental authority of the patients concerned by the research
* Malignant or benign solid tumor
* Thoracic, abdominal or pelvic location
* Clinico-radiological or histological diagnosis confirmed postnatally up to 1 year of life with onset of symptoms in the first three months of life
* Mother-child whose care course for the child's congenital axial tumor included treatment at the AP-HP

Exclusion Criteria:

* Opposition from holders of parental authority of patients
* Sacrococcygeal teratomas
* Central nervous system tumors
* Heart tumors
* Ovarian cysts
* Head and neck tumors
* Congenital leukemia and hemopathy

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mother-child whose care course for the child's congenital axial tumor included treatment at the AP-HP (Assistance Publique - Hôpitaux de Paris) between 2010 and 2021. Fetus presenting a malignant or benign solid tumor of thoracic, abdominal or pelvic location and whose clinico-radiological or histological diagnosis is confirmed postnatally up to 1 year of life with the onset of symptoms in the first three months of life.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Correlation between antenatal clinico-radiological analysis and postnatal diagnosis of solid congenital truncal tumors | 3 years
  Study of data from the patient's medical file.
Description of the developmental spectrum of solid congenital truncal tumors | 3 years
  Study of data from the patient's medical file.

SECONDARY OUTCOMES:
Characteristics and location of the tumor on pre- and post-natal imaging | 3 years
  Description of the characteristics and location of the tumor on pre- and post-natal imaging: ultrasound, MRI, CT scan.
Ile-de-France epidemiology of perinatal tumors | Through study completion, an average of 4 months
  Description of the epidemiology of perinatal tumors in the Paris region.
Evolution of solid congenital truncal tumors | Through study completion, an average of 4 months
  Description of the evolution of solid congenital truncal tumors.
Associated genetic abnormalities and malformations | Through study completion, an average of 4 months
  Description of genetic abnormalities and malformations that have been identified and associated with the tumor.
Intercurrent obstetric events and obstetric outcomes based on the diagnoses made | Through study completion, an average of 4 months
  Description of intercurrent obstetric events as well as the obstetric outcome based on the diagnoses made.
Development of a management algorithm based on prenatal findings | Through study completion, an average of 4 months
  Propose a management algorithm based on prenatal findings developed from the study data.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine SARNACKI, M.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Chelsea KHAWAND, M.D., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris

REFERENCES:
- [Background] Khawand C, Orbach D, Berrebi D, Branchereau S, Mussini C, Brisse HJ, Grevent D, Jouannic JM, Vivanti A, Minard-Colin V, Ville Y, Sarnacki S; Collaborators. Prenatal diagnosis and postnatal management of perinatal thoracoabdominopelvic tumors: multicenter experience. Ultrasound Obstet Gynecol. 2025 Oct;66(4):499-508. doi: 10.1002/uog.70000. Epub 2025 Aug 23. PMID 40847681
- [Background] Isaacs H Jr. Perinatal (congenital and neonatal) neoplasms: a report of 110 cases. Pediatr Pathol. 1985;3(2-4):165-216. doi: 10.3109/15513818509078782. PMID 3879355
- [Background] Moore SW, Satge D, Sasco AJ, Zimmermann A, Plaschkes J. The epidemiology of neonatal tumours. Report of an international working group. Pediatr Surg Int. 2003 Sep;19(7):509-19. doi: 10.1007/s00383-003-1048-8. Epub 2003 Sep 11. PMID 14523568
- [Background] Geurten C, Geurten M, Rigo V, Dresse MF. Neonatal Cancer Epidemiology and Outcome: A Retrospective Study. J Pediatr Hematol Oncol. 2020 Jul;42(5):e286-e292. doi: 10.1097/MPH.0000000000001692. PMID 31815889
- [Background] Parkes SE, Muir KR, Southern L, Cameron AH, Darbyshire PJ, Stevens MC. Neonatal tumours: a thirty-year population-based study. Med Pediatr Oncol. 1994;22(5):309-17. doi: 10.1002/mpo.2950220503. PMID 8127254
- [Background] Alamo L, Beck-Popovic M, Gudinchet F, Meuli R. Congenital tumors: imaging when life just begins. Insights Imaging. 2011 Jun;2(3):297-308. doi: 10.1007/s13244-011-0073-8. Epub 2011 Feb 14. PMID 22347954
- [Background] Avni FE, Massez A, Cassart M. Tumours of the fetal body: a review. Pediatr Radiol. 2009 Nov;39(11):1147-57. doi: 10.1007/s00247-009-1160-6. Epub 2009 Feb 24. PMID 19238373
- [Background] Orbach D, Sarnacki S, Brisse HJ, Gauthier-Villars M, Jarreau PH, Tsatsaris V, Baruchel A, Zerah M, Seigneur E, Peuchmaur M, Doz F. Neonatal cancer. Lancet Oncol. 2013 Dec;14(13):e609-20. doi: 10.1016/S1470-2045(13)70236-5. PMID 24275134
- [Background] Kamil D, Tepelmann J, Berg C, Heep A, Axt-Fliedner R, Gembruch U, Geipel A. Spectrum and outcome of prenatally diagnosed fetal tumors. Ultrasound Obstet Gynecol. 2008 Mar;31(3):296-302. doi: 10.1002/uog.5260. PMID 18307207
- [Background] Amari F, Beyer DA, Diedrich K, Weichert J. Fetal intra-abdominal tumors: assessment of spectrum, accuracy of prenatal diagnosis, perinatal outcome and therapy at a tertiary referral center. Eur J Obstet Gynecol Reprod Biol. 2013 Apr;167(2):160-6. doi: 10.1016/j.ejogrb.2012.11.023. Epub 2013 Jan 5. PMID 23295072
- [Background] Meizner I. Perinatal oncology--the role of prenatal ultrasound diagnosis. Ultrasound Obstet Gynecol. 2000 Nov;16(6):507-9. doi: 10.1046/j.1469-0705.2000.00297.x. No abstract available. PMID 11169341
- [Background] Isaacs H Jr. Fetal hydrops associated with tumors. Am J Perinatol. 2008 Jan;25(1):43-68. doi: 10.1055/s-2007-1004826. Epub 2007 Dec 12. PMID 18075961
- [Background] Braun T, Brauer M, Fuchs I, Czernik C, Dudenhausen JW, Henrich W, Sarioglu N. Mirror syndrome: a systematic review of fetal associated conditions, maternal presentation and perinatal outcome. Fetal Diagn Ther. 2010;27(4):191-203. doi: 10.1159/000305096. Epub 2010 Mar 27. PMID 20357423
- [Background] Sauvat F, Sarnacki S, Brisse H, Medioni J, Rubie H, Aigrain Y, Gauthier F, Audry G, Helardot P, Landais P, Michon J, Hartmann O, Nihoul-Fekete C. Outcome of suprarenal localized masses diagnosed during the perinatal period: a retrospective multicenter study. Cancer. 2002 May 1;94(9):2474-80. doi: 10.1002/cncr.10502. PMID 12015773